CLINICAL TRIAL: NCT06911281
Title: Clinical Study on the Combination Therapy of Photoelectric Instruments and Human Umbilical Cord Mesenchymal Stem Cells for Pigmentary Disorders
Brief Title: Combined Therapy of Photoelectric Instruments and Human Umbilical Cord Mesenchymal Stem Cells for Pigmentary Disorders
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: ARSMO(Hainan) International Plastic & Aesthetic Hospital Company Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFSC-2025(CR)-01
Record Dates: First submitted 2025-03-23; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Mesenchymal Stem Cells；Pigmentary Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stem Cell Treatment Group 1 (Experimental): Administer MSCs via intravenous infusion and multi-point injection into the melasma area, followed by combined treatment with 755nm picosecond laser.
  Interventions: Combination Product: Mesenchymal Stem Cells；755nm picosecond laser treatment
- Stem Cell Treatment Group 2 (Experimental): Administer MSCs via multi-point injection into the melasma area, followed by combined treatment with 755nm picosecond laser.
  Interventions: Combination Product: Mesenchymal Stem Cells；755nm picosecond laser treatment
- Control Group (Experimental): Only administer 755nm picosecond laser treatment.
  Interventions: Combination Product: Mesenchymal Stem Cells；755nm picosecond laser treatment

INTERVENTIONS:
Combination Product: Mesenchymal Stem Cells；755nm picosecond laser treatment — Stem Cell Treatment Group 1 received intravenous infusion of MSCs followed by multi-point injection into the melasma area, combined with 755nm picosecond laser treatment. Stem Cell Treatment Group 2 received multi-point injection of MSCs into the melasma area, combined with 755nm picosecond laser treatment. The Control Group only received 755nm picosecond laser treatment.

SUMMARY:
Melasma is a common and refractory pigmentary skin disorder manifested as light to dark brown patches on the facial skin. It belongs to disfiguring dermatoses and significantly affects the physical and mental well-being of patients. Conventional treatments for melasma, including pharmacological and photoelectric therapies, have high recurrence rates and suboptimal clinical efficacy. Preliminary evaluations of the therapeutic effects of human umbilical cord mesenchymal stem cells (MSCs) in melasma mouse models have shown that MSCs can significantly improve skin pigmentation, reduce malondialdehyde (MDA) levels indicating anti-aging effects, ameliorate skin inflammatory cell infiltration, and promote skin repair in these models. This study is a single-center, randomized controlled clinical trial aiming to build on previous experimental findings by combining MSCs with photoelectric therapy for the treatment of melasma. Patients will be divided into three groups of 10 each: Stem Cell Treatment Group 1, Stem Cell Treatment Group 2, and a Control Group. Group 1 will receive intravenous infusion of MSCs followed by multi-point injection into the melasma area in combination with 755nm picosecond laser treatment. Group 2 will receive multi-point injection of MSCs into the melasma area in combination with 755nm picosecond laser treatment. The Control Group will only receive 755nm picosecond laser treatment. Efficacy will be initially assessed based on parameters such as the Melasma Area and Severity Index (MASI), VISIA skin analysis, and patient satisfaction. The study aims to evaluate the efficacy and safety of MSCs combined with photoelectric therapy for melasma and to investigate the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily participate in this study and sign a written informed consent form.
2. Subjects are female patients with melasma aged between 18 and 60 years. Their diagnosis should conform to the "Chinese Expert Consensus on Diagnosis and Treatment of Melasma (2021 Edition)" formulated by the Pigmentary Disorders Subgroup of the Dermatovenereology Committee of the China Association of Integrative Medicine. The skin lesions manifest as light brown or dark brown patches of varying depths and with indistinct borders on the cheeks, forehead, and jaw. Subjects must be excluded from having post-inflammatory hyperpigmentation, naevus of Ota, Riehl's melanosis, pigmented lichen planus, and other skin diseases. Additionally, their melasma should have been in a stable phase for 3 months or more.
3. Subjects have never undergone stem cell therapy or laser treatment for melasma.

Exclusion Criteria:

1. Subjects with a history of photosensitivity or allergies to biological medications.
2. Subjects who are pregnant or lactating.
3. Subjects who have a history of alcohol abuse, drug addiction, or substance abuse in the past 24 months.
4. Subjects with concurrent severe systemic diseases, malignancies, or psychiatric disorders.
5. Subjects with active infections, including bacterial, fungal, and viral infections.
6. Subjects with keloid constitution.
7. Subjects with a history of severe sun exposure within 4 weeks before enrollment.
8. Subjects deemed unsuitable for enrollment by the investigator for various reasons or any other conditions that the investigator believes may compromise the safety or compliance of the subject or hinder the successful completion of the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation endpoint | From 0 days to 2 years
  The number of adverse events occurring throughout the entire study period. Analyze the frequency and occurrence of adverse events (including injection site reactions). Calculate adverse events, adverse reactions, and AE causing detachment separately SAE、 The number and frequency of AE with different degrees of severity and AE causing death.
  Secondary endpoints: The primary evaluation includes the therapeutic effect of melasma and local discomfort.
Pigmented Disease Area and Severity Index (MASI) | From 0 days to 2 years
  Quantitative analysis based on the area, depth, and uniformity of pigmentary diseases. Assess pigmentation areas in four regions: forehead (F) 30%, right cheek (MR) 30%, left cheek (ML) 30%, and mandible (C) 10%. According to the proportion of pigmentation spots in the four regions, the scores are: 1 is less than 10%, 2 is 10% -29%, 3 is 30% -49%, 4 is 50% -69%, 5 is 70% -89%, and 6 is 90% -100%. Color depth (D) and uniformity (H) scores: 0-4 points: none 0 points, slight 1 point, moderate 2 points, obvious 3 points, highest 4 points. MASI=forehead [0.3A (D+H)]+right cheek [0.3A (D+H)]+left cheek [0.3A (D+H)]+mandible [0.1A (D+H)]. The highest score is 48 points, and the lowest score is 0 points.
VISIA Image Analysis System | From 0 days to 2 years
  VISIA image analysis system: uses different light sources such as standard, ultraviolet, and orthogonal polarization to quantify different skin states. Patients with pigmentary diseases can determine the quantity, distribution, area, depth, and capillary condition of pigments through surface, ultraviolet, and brown spots.

IPD SHARING:
Plan to Share IPD: No